CLINICAL TRIAL: NCT06957990
Title: Evaluation of Music Therapy for Pre-op/Intra-op During Hernia Surgery to Decrease the Need for Narcotics
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 24-060
Record Dates: First submitted 2025-04-21; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Surgery; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Preoperative music will be unmasked. Intraoperative music will be masked - Only research nurse will know if music was turned on or off intraoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PreOp Only (Experimental): Patient will listen to music before their surgery in pre-operative area only
  Interventions: Other: Music
- PreOp and IntraOp (Experimental): Patient will listen to music before and during their surgery
  Interventions: Other: Music
- IntraOp Only (Experimental): Patient will listen to music during their surgery only
  Interventions: Other: Music
- No Music (No Intervention): Patient will not listen to music during their visit

INTERVENTIONS:
Other: Music — Music of the participant's selected genre will be played through headphones according to the arm assigned.
  Arms: IntraOp Only; PreOp Only; PreOp and IntraOp

SUMMARY:
The purpose of this study is to investigate if audible distraction, in the form of music, before and/or during hernia repair surgery will decrease pain post-operatively.

DETAILED DESCRIPTION:
After performing a thorough review of the literature, no studies were found that examined whether having a patient listen to a genre of music of their choosing before or during surgery impacts their postoperative pain. Music is a way to relax patients and could potentially decrease pain, which is a goal of perioperative services. The current study seeks to fill the gap and examine the impact of music on pain for surgical patients undergoing a hernia repair.

This study will use a randomized, double-blinded, controlled design with four arms:

* Arm 1: Patient will listen to music before their surgery in pre-operative area only
* Arm 2: Patient will listen to music before and during their surgery
* Arm 3: Patient will listen to music during their surgery only
* Arm 4: Patient will not listen to music during their visit

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Receiving surgery at Bethesda Surgery Center

Exclusion Criteria:

* Does not speak English
* Unable to consent to involvement in the research study
* Having more than 1 hernia repair performed
* Pregnant
* Deaf
* Wears hearing aids
* Currently on medication-assisted treatment for substance use disorder (ex: suboxone or methadone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-08-08 (Estimated); Study Completion 2026-10-08 (Estimated)

PRIMARY OUTCOMES:
Highest pain score reported | from admission to discharge from PACU, up to 8 hours
  Highest pain score reported in the Post Anesthesia Care Unit (PACU); Pain is measured on a 0-10 scale where a higher number corresponds with more pain
Total narcotic administered | from admission to discharge from PACU, up to 8 hours
  Total morphine milligram equivalent (MME) of narcotics administered while in PACU

CONTACTS AND LOCATIONS:
Locations (1):
- Bethesda Surgery Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No